CLINICAL TRIAL: NCT02714985
Title: RT-PCR on Urine Samples: Added Value for the Diagnosis of Chikungunya Virus Infection
Acronym: CHIK_urine
Status: Withdrawn | Type: Observational
Why Stopped: not able to recruit participants
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: B300201525794
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Chikungunya Fever
Keywords: chikungunya virus; RT-PCR; urine; diagnosis
MeSH Terms: conditions — Chikungunya Fever; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- confirmed chikungunya cases: cases with confirmed chikungunya fever and included for follow-up as per protocol

SUMMARY:
Retrospective laboratory evaluation of the detection rate of CHIKV infection by real-time Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) on urine. Urine and serum samples from patients with confirmed CHIKV infections from an endemic area (Aruba) and from ITM will be analyzed. The results will be evaluated on a case-by-case basis: time since onset, patient characteristics, severity of symptoms, serology results.

The positivity in-time of CHIKV RNA in urine will be evaluated in comparison with viremia. Patients with suspected acute CHIKV infection will be asked (by written informed consent; annex 1) to provide urine samples within 72 hours after onset of disease, followed by urine samples on day 7, day 10, day 14 and three urine samples 3, 4 and 12 weeks after onset. They will be asked to provide serum samples within 72 hours after onset of disease, followed by serum samples on day 7, day 10, day 14. In total, twenty patients with an initial positive result of CHIKV RT-PCR on serum will be included for follow-up. The number of urine samples that will be tested is 140.

DETAILED DESCRIPTION:
Objectives

1. To assess the added value of RT-PCR for CHIKV on urine samples for diagnosing CHIKV infection in comparison to the reference methods.
2. To describe the kinetics of RT- PCR for CHIKV on urine samples for diagnosing CHIKV infection over time.

Study design, population, materials and methods:

Prospective cohort study of patients with a confirmed CHIKV infection (positive RT-PCR for CHIKV on the sample at the time of inclusion or seroconversion defined as positive anti-CHIKV Immunoglobulin M (IgM) antibody assay on day 14), who attend the outpatient clinic of the Institute of Tropical Medicine in Antwerp and the Horacio Oduber Hospitaal in Aruba within 72 hours after fever onset. After signing informed consent, clinical and epidemiological data will be recorded in a standardized Case Record Form. Baseline blood and urine samples will be collected as required for routine clinical evaluation of the individual case; sampling will include serum CHIKV serologic assays, CHIKV E1 (or similar rapid test), as well as serum and urine for RT-PCR for CHIKV. After the initial evaluation, suspected CHIKV cases are scheduled for biweekly serum and urine collection for RT-PCR for CHIKV for a duration of 2 weeks, then after 3, 4 and 12 weeks. Serum at 4 weeks will be used for second serologic assay. Suspected cases that test negative for CHIKV by RT-PCR on serum will be excluded.

Study population : patients with confirmed CHIKV infection Sample size : panel of 20 CHIKV confirmed cases Data analysis and reporting : The percentages of positive urine RT-PCR (over different time-points of duration of the CHIKV infection) will be calculated. Proportions of positivity rates will be tested by χ²-test for equality of proportions. Ct-values between two different sample types (serum/urine) will be compared by calculation of Spearman's rank correlation coefficient (ρ). The Ct-values measured will be subtracted (indicated by ∆Ct) and the mean of all ∆Ct-values (± 95% confidence interval) will be calculated. Reporting in accordance with Standards for Reporting of Diagnostic Accuracy (STARD) guidelines.

Endpoints: diagnostic sensitivity of CHIKV RT-PCR on urine samples in patients with a confirmed CHIKV infection, comparison of analytical sensitivity (based on Ct-values) with RT-PCR on serum, positivity rates of RT-PCR urine samples over time Ethical issues: Informed consent will be obtained from study participants. Demographic, geographic, clinical and laboratory data will be obtained; the data are de-identified and stored in an encoded database (code known to the principal investigators). Ethical approval through the ITM/ University Hospital Antwerp (UZA) Ethics Committee (EC) and the EC in Aruba.

Expected results and relevance :

Evaluation of the sensitivity of RT-PCR on urine samples for diagnosing CHIKV infection in the post-viremic phase in both endemic and non-endemic settings. Possible advantages of the use of PCR on urine over serological assays are:

1. a shift in timeframe for accurately diagnosing CHIKV infection that could benefit returning travelers who consult after the acute phase.
2. the use of single specimens that are obtained by non-invasive procedures
3. high specificity
4. the opportunity for typing of CHIKV strains.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* clinical suspicion of CHIKV infection, i.e.
* fever (≥38°C) AND arthralgia OR rash
* Confirmation of CHIKV infection by RT-PCR on serum or seroconversion (defined as positive anti-CHIKV IgM antibody assay on day 14)
* living within 50 kilometer of either study site (ITM Antwerp, on Aruba)
* Willing and able to provide written informed consent (assent for minors).

Exclusion Criteria:

* Alternative diagnosis at the time of evaluation
* Unable to produce urine sample by spontaneous micturition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a confirmed chikungunya virus (CHIKV) infection, who attend the outpatient clinic of the Institute of Tropical Medicine in Antwerp or the Horacio Oduber Hospitaal in Aruba within 72 hours after fever onset.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
detection rate of chikungunya virus by RT-PCR in urine samples | 12 weeks
  in patients with a confirmed CHIKV infection, comparison of analytical sensitivity (based on Ct-values) with RT-PCR on serum, positivity rates of RT-PCR urine samples over time

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, MD PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium
Locations (2):
- Horacio Oduber Hospitaal, Oranjestad, Aruba
- ITM, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barzon L, Pacenti M, Franchin E, Pagni S, Martello T, Cattai M, Cusinato R, Palu G. Excretion of West Nile virus in urine during acute infection. J Infect Dis. 2013 Oct 1;208(7):1086-92. doi: 10.1093/infdis/jit290. Epub 2013 Jul 2. PMID 23821721
- [Background] Blacksell SD, Tanganuchitcharnchai A, Jarman RG, Gibbons RV, Paris DH, Bailey MS, Day NP, Premaratna R, Lalloo DG, de Silva HJ. Poor diagnostic accuracy of commercial antibody-based assays for the diagnosis of acute Chikungunya infection. Clin Vaccine Immunol. 2011 Oct;18(10):1773-5. doi: 10.1128/CVI.05288-11. Epub 2011 Aug 24. PMID 21865416
- [Background] Couturier E, Guillemin F, Mura M, Leon L, Virion JM, Letort MJ, De Valk H, Simon F, Vaillant V. Impaired quality of life after chikungunya virus infection: a 2-year follow-up study. Rheumatology (Oxford). 2012 Jul;51(7):1315-22. doi: 10.1093/rheumatology/kes015. Epub 2012 Mar 16. PMID 22427407
- [Background] Gourinat AC, O'Connor O, Calvez E, Goarant C, Dupont-Rouzeyrol M. Detection of Zika virus in urine. Emerg Infect Dis. 2015 Jan;21(1):84-6. doi: 10.3201/eid2101.140894. PMID 25530324
- [Background] Hirayama T, Mizuno Y, Takeshita N, Kotaki A, Tajima S, Omatsu T, Sano K, Kurane I, Takasaki T. Detection of dengue virus genome in urine by real-time reverse transcriptase PCR: a laboratory diagnostic method useful after disappearance of the genome in serum. J Clin Microbiol. 2012 Jun;50(6):2047-52. doi: 10.1128/JCM.06557-11. Epub 2012 Mar 21. PMID 22442323
- [Background] Korhonen EM, Huhtamo E, Virtala AM, Kantele A, Vapalahti O. Approach to non-invasive sampling in dengue diagnostics: exploring virus and NS1 antigen detection in saliva and urine of travelers with dengue. J Clin Virol. 2014 Nov;61(3):353-8. doi: 10.1016/j.jcv.2014.08.021. Epub 2014 Sep 1. PMID 25242312
- [Background] Magurano F, Zammarchi L, Baggieri M, Fortuna C, Farese A, Benedetti E, Fiorentini C, Rezza G, Nicoletti L, Bartoloni A. Chikungunya from the Caribbean: the importance of appropriate laboratory tests to confirm the diagnosis. Vector Borne Zoonotic Dis. 2015 Apr;15(4):258-60. doi: 10.1089/vbz.2014.1724. PMID 25897812
- [Background] Mizuno Y, Kotaki A, Harada F, Tajima S, Kurane I, Takasaki T. Confirmation of dengue virus infection by detection of dengue virus type 1 genome in urine and saliva but not in plasma. Trans R Soc Trop Med Hyg. 2007 Jul;101(7):738-9. doi: 10.1016/j.trstmh.2007.02.007. Epub 2007 Apr 5. PMID 17418320
- [Background] Panning M, Grywna K, van Esbroeck M, Emmerich P, Drosten C. Chikungunya fever in travelers returning to Europe from the Indian Ocean region, 2006. Emerg Infect Dis. 2008 Mar;14(3):416-22. doi: 10.3201/eid1403.070906. PMID 18325256
- [Background] Van den Bossche D, Cnops L, Van Esbroeck M. Recovery of dengue virus from urine samples by real-time RT-PCR. Eur J Clin Microbiol Infect Dis. 2015 Jul;34(7):1361-7. doi: 10.1007/s10096-015-2359-0. Epub 2015 Mar 21. PMID 25794553